CLINICAL TRIAL: NCT00586898
Title: Rapid Hormonal Cycling as Treatment for Patients With Prostate Cancer: The Men's Cycle
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-085
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Prostate; Cancer; Hormonal Cycling
Keywords: Prostate; Cancer; Hormones; 01-085; ANTIFUNGAL ANTIBIOTICS; ESTROGENS; LUPRON; TESTOSTERONE; ZOLADEX
MeSH Terms: conditions — Neoplasms | interventions — Gonadotropin-Releasing Hormone; Leuprolide; Goserelin; Ketoconazole; bicalutamide; Testosterone; Estradiol

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GnRH; Drug: Ketoconazole; Drug: Bicalutamide; Drug: Testosterone transdermal gel; Drug: Estrogen transdermal patch

INTERVENTIONS:
Drug: GnRH — leuprolide and goserelin are gonadotropin-releasing hormone analogues
  Other Names: LUPRON; ZOLADEX
Drug: Ketoconazole — An imidazole antifungal agent. reduces adrenal and testicular androgen production in men
  Other Names: Nizoral
Drug: Bicalutamide — A pure nonsteroidal antiandrogen
  Other Names: Casodex
Drug: Testosterone transdermal gel — an androgenic anabolic steroid
  Other Names: Androgel
Drug: Estrogen transdermal patch — Estradiol is the primary and most potent estrogen
  Other Names: CLIMARA

SUMMARY:
Objective: To determine the response to rapid hormonal cycling in patients with non-castrate prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

-Patients residing in the following clinical states wit! be considered: A. Rising PSA: Patients with a history of localized disease who have undergone definitive radiation or surgery. These patients must demonstrate progression of disease biochemically as outlined below. Patients in this group may not have radiographically evident disease.

B. Non-castrate metastatic: Patients must present with radiographic evidence of metastatic disease at the time of diagnosis or after treatment for localized disease. These patients must show newly detected disease or progressing disease in bone or in soft tissue. Biochemical progression is defined as: minimum no. of determinations: 3 Interval: >2 weeks Minimal Baseline PSA value (ng/ml): 2 Minimal % increase in range of values: 50%

* Diagnosis of prostate adenocarcinoma histologically confirmed at MSKCC.
* Patient must have level of serum testosterone above the lower limit of normal.
* Karnofskcy performance status (KPS) >_70%.
* Patients must have adequate organ function as defined by the following laboratory criteria:
* WBC >_3500/mm3, platelet count >_100,000/mm3.
* Bilirubin <2.0 mg/dl or SGOT <3.0 X the upper limit of normal.
* Creatinine <_1.6 mg/dl or creatinine clearance >_60 cc/min.
* Prior hormonal therapy is allowed as:

  1. Neoadjuvant treatment prior to radiation therapy or radical prostatectomy, provided that the total duration of exposure does not exceed 10 months.
  2. One cycle of intermittent therapy up to a maximum exposure of 10 months.
* Patients must be at least 18 years of age.
* Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment

Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III/IV),or severe debilitating puhnonary disease.
* Uncontrolled serious active infection.
* Anticipated survival of less than 3 months.
* Active CNS or epiduraltumor
* Inability or unwillingness to comply with the treatment protocol, follow-up, or research tests.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2001-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Scher, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Rapid Hormonal Cycling as Treatment for Patients with Prostate Cancer
Period: Overall Study
Arm/Group | All Participants
Started | 36
Completed | 29
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Patiemt Non-compliance | 1
Not completed — Evaluable for Toxicity Only | 5

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Complete Response: Normalization of the PSA (< or = to 4.0 for patients with castrate metastatic disease, or < 0.5 for patients with a rising PSA) that is maintained on 3 successive evaluations a minimum of 2 weeks apart. Partial Response: Decrease in PSA value by > or = to 50% from baseline value (without normalization) for 3 successive evaluations a minimum of 2 weeks apart. Stabilization: Patients who do not meet the criteria for PR or PROG for at least 90 days will be considered stable.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 29
participants
  Complete Response (CR) | 22
  Partial Response (PR) | 4
  Stable Disease (SD) | 3

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 2/36
Other Adverse Events (participants affected / at risk) | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=36)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiovascular, other (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hot Flashes (General disorders) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
SGPT (ALT) (Metabolism and nutrition disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes